CLINICAL TRIAL: NCT03352453
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Efficacy and Safety Study of Rapastinel for Rapid Treatment of Symptoms of Depression and Suicidality in Adult Patients With Major Depressive Disorder
Brief Title: A Study of Rapastinel for Rapid Treatment of Depression and Suicidality in Major Depressive Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped due to business reasons.
Sponsor: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAP-MD-20
Record Dates: First submitted 2017-11-21; First posted 2017-11-24 (Actual); Results first posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-07

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — GLYX-13 peptide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rapastinel 450mg (Experimental): Rapastinel 450 milligram (mg) weekly intravenous (IV) injections.
  Interventions: Drug: Rapastinel
- Placebo (Placebo Comparator): Placebo-matching rapastinel weekly IV injections.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rapastinel — Rapastinel pre-filled syringes for weekly IV injections.
  Arms: Rapastinel 450mg
Drug: Placebo — Placebo-matching rapastinel pre-filled syringes for weekly IV injections.
  Arms: Placebo

SUMMARY:
The study will evaluate the efficacy, safety, and tolerability of 450 milligrams (mg) of Rapastinel, compared to placebo in adult patients with major depressive disorder (MDD) who are at imminent risk of suicide.

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) criteria for MDD
* Current major Depressive episode of at least 4 weeks and not exceeding 24 months in duration at visit 1
* Have current, ongoing suicidality (ideation or behavior) of sufficient severity to warrant hospitalization based on the judgment of the investigator
* If female of childbearing potential, have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test.

Exclusion Criteria:

* DSM-5-based diagnosis of any disorder other than MDD that was the primary focus of treatment within 1 month before Visit 1.
* Lifetime history or currently meet DSM-5 criteria for:

  1. Schizophrenia spectrum or other psychotic disorder
  2. Bipolar or related disorder
  3. Major neurocognitive disorder
  4. Neurodevelopmental disorder of greater than mild severity or of a severity that impacts the participant's ability to consent, follow study directions, or otherwise safely participate in the study.
  5. Dissociative disorder
  6. Posttraumatic stress disorder
  7. MDD with psychotic features
* Significant homicidal ideation or at imminent risk of injuring others or causing significant damage to property, as judged by the investigator.
* Prior participation in any investigational study of rapastinel/GLYX-13

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Hoogerheyde, Study Director — Allergan
Locations (17):
- United States (17):
  - The Board of Trustees of the University of Alabama for the University of Alabama at Birmingham, Birmingham, Alabama
  - Collaborative NeuroScience Network, LLC, Garden Grove, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Asclepes Research Centers, Panorama City, California
  - Institute of Living, Hartford, Connecticut
  - Innovative Clinical Research, Inc, Hialeah, Florida
  - Research Centers of America, LLC, Oakland Park, Florida
  - Atlanta Center for Medical Research (ACMR), Atlanta, Georgia
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - CBH Health, Gaithersburg, Maryland
  - Altea Research Institute, Las Vegas, Nevada
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - Pillar Clinical Research, LLC, Richardson, Texas
  - Carilion Medical Center, a Virginia Nonprofit Corporation, Roanoke, Virginia
  - Department of Veterans Affairs Salem VA Medical Center, Salem, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance. — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Rapastinel 450mg
Started | 66 | 72
Completed | 44 | 40
Not Completed | 22 | 32
Not completed — Miscellaneous Reasons | 1 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 8 | 14
Not completed — Study Terminated by Sponsor | 2 | 1
Not completed — Protocol Deviation | 1 | 0
Not completed — Lost to Follow-up | 7 | 6
Not completed — Adverse Event | 2 | 9

BASELINE CHARACTERISTICS:
Population: The modified Intent-to-Treat (mITT) Population will consist of all patients in the Safety Population who had at least 1 postbaseline assessment of the MADRS total score or S-STS total score.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rapastinel 450mg | Total
Number analyzed (Participants) | 64 | 72 | 136
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.1 (13.45) | 42.3 (12.89) | 42.2 (13.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 35 | 43 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 11 | 20
  Not Hispanic or Latino | 55 | 61 | 116
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 33 | 24 | 57
  White | 30 | 45 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Montgomery-Asberg Depression Rating Scale (MADRS) total score at baseline [Mean (Standard Deviation); unit: Scores on a scale] — The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. Participants are rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and a lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score ranges from 0 to 60 with a higher score indicating more depression.
  Scores on a scale | 40.4 (5.83) | 39.8 (6.04) | 40.0 (5.93)
Sheehan - Suicidality Tracking Scale (S-STS) Total Score (Patient-rated) [Mean (Standard Deviation); unit: Scores on a scale] — The S-STS is a patient-report informed, clinician-rated scale used to rate the severity of suicidal impulses, thoughts, and behaviors. This is a 14 item scale ranging from 0=Not at all to 4= Extremely. The total score ranges from 0 to 56 with a higher score indicating higher suicidal tendency.
  Scores on a scale | 30.9 (10.94) | 29.6 (10.45) | 30.2 (10.67)
Weight [Mean (Standard Deviation); unit: kg] | 85.26 (19.80) | 82.57 (17.59) | 83.83 (18.64)
Height [Mean (Standard Deviation); unit: cm] | 172 (8.84) | 169.56 (9.86) | 170.71 (9.44)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.88 (6.75) | 28.79 (6.34) | 28.83 (6.51)
S-STS Total Score (Clinician-rated) [Mean (Standard Deviation); unit: Scores on a scale] — The S-STS is a patient-report informed, clinician-rated scale used to rate the severity of suicidal impulses, thoughts, and behaviors. This is a 14 item scale ranging from 0=Not at all to 4= Extremely. The total score ranges from 0 to 56 with a higher score indicating higher suicidal tendency.
  Scores on a scale | 30.0 (10.22) | 28.9 (9.62) | 29.4 (9.88)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. Participants are rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and a lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score ranges from 0 to 60 with a higher score indicating more depression. A negative change score indicates improvement.
Time Frame: Baseline and 1 Day
Population: The modified Intent-to-Treat (mITT) Population consists of all participants in the Safety Population who had at least 1 postbaseline assessment of the MADRS total score or S-STS total score.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Rapastinel 450mg
Number analyzed (Participants) | 64 | 72
Scores on a scale | -17.6 (12.49) | -16.3 (11.36)

2. Primary Outcome: Change From Baseline in Sheehan - Suicidality Tracking Scale (S-STS) Total Score
Description: The S-STS is a patient-report informed, clinician-rated scale used to rate the severity of suicidal impulses, thoughts, and behaviors. This is a 14 item scale ranging from 0=Not at all to 4= Extremely. The total score ranges from 0 to 56 with a higher score indicating higher suicidal tendency.
Time Frame: Baseline and 1 Day
Population: The modified Intent-to-Treat (mITT) Population consists of all patients in the Safety Population who had at least 1 postbaseline assessment of the MADRS total score or S-STS total score.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Rapastinel 450mg
Number analyzed (Participants) | 64 | 72
Scores on a scale | -20.6 (12.27) | -20.2 (11.93)

3. Secondary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: as for outcome 1
Time Frame: Baseline and 28 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Rapastinel 450mg
Number analyzed (Participants) | 64 | 72
Scores on a scale | -25.6 (14.74) | -23.0 (15.00)

4. Secondary Outcome: Change From Baseline in Sheehan - Suicidality Tracking Scale (S-STS) Total Score
Description: as for outcome 2
Time Frame: Baseline and 28 Days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Rapastinel 450mg
Number analyzed (Participants) | 64 | 72
Scores on a scale | -25.9 (11.61) | -26.4 (12.74)

ADVERSE EVENTS:
Time Frame: The study consisted of a 4 week double-blind treatment period, followed by a 1-week safety follow-up period.
Description: The Safety Population will consist of all patients in the Randomized Population who took at least 1 dose of randomized IP.
Arm/Group | Placebo | Rapastinel 450mg
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/72
Serious Adverse Events (participants affected / at risk) | 5/64 | 12/72
Other Adverse Events (participants affected / at risk) | 18/64 | 21/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=64) | Rapastinel 450mg (N=72)
Suicidal ideation (Psychiatric disorders) | 3 | 5
Non-cardiac chest pain (General disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Depressive Symptom (Psychiatric disorders) | 1 | 1
Suicide attempt (Psychiatric disorders) | 0 | 3
Major Depression (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Mitral Valve Incompetence (Cardiac disorders) | 0 | 1
Mitral Valve Prolapse (Cardiac disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=64) | Rapastinel 450mg (N=72)
Anxiety (Psychiatric disorders) | 5 | 5
Headache (Nervous system disorders) | 5 | 6
Insomnia (Psychiatric disorders) | 3 | 6
Dizziness (Nervous system disorders) | 3 | 5
Nausea (Gastrointestinal disorders) | 5 | 4

LIMITATIONS AND CAVEATS:
Due to study termination, the target number of participants needed to achieve target power and statistically reliable results was not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT03352453/SAP_000.pdf
  • Study Protocol (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT03352453/Prot_001.pdf